CLINICAL TRIAL: NCT00828009
Title: A Phase II Study of L-BLP25 and Bevacizumab in Unresectable Stage IIIA and IIIB Non-Squamous Non-Small Cell Lung Cancer After Definitive Chemoradiation
Brief Title: BLP25 Liposome Vaccine and Bevacizumab After Chemotherapy and Radiation Therapy in Treating Patients With Newly Diagnosed Stage IIIA or Stage IIIB Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000632611; E6508 (Other: ECOG-ACRIN Cancer Research Group); U10CA180794 (NIH)
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Bevacizumab; L-BLP25; Carboplatin; Cyclophosphamide; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tecemotide/bevacizumab after chemoradiation (Experimental): Concomitant Chemoradiotherapy: Patients (pts) receive paclitaxel intravenously (IV) over 1 hour and carboplatin IV over 15-30 minutes weekly for 6 weeks. Pts also receive radiotherapy 5 days a week for 6½ weeks. Pts with CR, PR, or SD proceed to consolidation chemotherapy.
  Consolidation chemotherapy: Pts receive paclitaxel IV over 3 hours and carboplatin IV over 15-30 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression (PD) or unacceptable toxicity. Pts with CR, PR, or SD proceed to maintenance therapy.
  Maintenance therapy: Pts receive a single dose of cyclophosphamide IV over 15-30 minutes 3 days before the first dose of bevacizumab and tecemotide. Pts then receive bevacizumab IV over 30-90 minutes on day 1 and tecemotide subcutaneously on days 1, 8, and 15 of courses 1 and 2 and on day 1 of every other course beginning in course 4. Treatment repeats every 21 days for up to 34 courses in the absence of PD or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Biological: Tecemotide; Drug: carboplatin; Drug: cyclophosphamide; Drug: paclitaxel; Radiation: radiotherapy

INTERVENTIONS:
Biological: bevacizumab — IV
  Other Names: NSC 704865; RhuMAb VEGF; Recombinant Humanized Monoclonal Bevacizumab Antibody
Biological: Tecemotide
  Other Names: L-BLP25
Drug: carboplatin — IV
  Other Names: CBDCA; paraplatin; JM-8; NSC 241240
Drug: cyclophosphamide — IV
  Other Names: Cytoxan; Neosar; CTX; CPM
Drug: paclitaxel — IV
  Other Names: taxol; NSC #673089
Radiation: radiotherapy — radiotherapy is given 5 days a week for 6½ weeks during concomitant chemoradiotherapy

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response to kill tumor cells. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving vaccine therapy together with bevacizumab after chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving BLP25 liposome vaccine together with bevacizumab after chemotherapy and radiation therapy in treating patients with newly diagnosed stage IIIA or stage IIIB non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety of BLP25 liposome vaccine (tecemotide) and bevacizumab after definitive chemoradiotherapy and consolidation chemotherapy in patients with newly diagnosed, unresectable stage IIIA or IIIB nonsquamous cell non-small cell lung cancer.

Secondary

* To evaluate the overall survival and progression-free in patients treated with this regimen.
* To evaluate the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Step 1:

* Chemoradiotherapy: Patients receive paclitaxel intravenously (IV) over 1 hour and carboplatin IV over 15-30 minutes once a week for 6 weeks. Patients also undergo concurrent definitive radiotherapy 5 days a week for 6½ weeks. Patients with complete response (CR), partial response (PR), or stable disease (SD) proceed to consolidation chemotherapy.
* Consolidation chemotherapy: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 15-30 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with CR, PR, or SD proceed to maintenance therapy.

Step 2:

* Maintenance therapy: Patients receive a single dose of cyclophosphamide IV over 15-30 minutes 3 days before the first dose of bevacizumab and BLP25 liposome vaccine. Patients then receive bevacizumab IV over 30-90 minutes on day 1 and BLP25 liposome vaccine subcutaneously on days 1, 8, and 15 of courses 1 and 2 and on day 1 of every other course beginning in course 4. Treatment repeats every 21 days for up to 34 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Step 1 Inclusion Criteria:

* Histologically confirmed newly diagnosed nonsquamous non-small cell lung cancer (NSCLC), including the following subtypes:

  * Adenocarcinoma
  * Large cell undifferentiated
  * Bronchoalveolar cell
  * non-small cell carcinoma, not otherwise specified
* Unresectable stage IIIA or stage IIIB disease

  * Patients with stage IIIA disease with mediastinal lymph node enlargement between 1 cm and 2.0 cm on computerized tomography (CT) scan must have these nodes biopsied (pathologic confirmation) to rule out resectability
  * Metastases to contralateral mediastinal or supraclavicular nodes allowed
* Measurable or non-measurable disease, as defined by Response Evaluation Criteria in Solid Tumours (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* White blood cell (WBC) ≥ 4,000/mm³ OR Absolute neutrophil count (ANC) ≥ 2,000/mm³
* Platelet count ≥ 140,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT)+ ≤ 2.5 times upper limit of normal
* Serum creatinine ≤ 1.5 mg/mL OR creatinine clearance ≥ 45 mL/min
* Urine protein:creatinine ratio < 1.0 by urine dipstick OR < 1 g of protein by 24-hour urine collection
* INR ≤ 1.5 OR ≤ 3.0 if patient is on therapeutic anticoagulation
* PTT normal
* Fertile patients must use effective contraception before, during, and for ≥ 6 months after completion of bevacizumab

Step 1 Exclusion Criteria:

* Significant pleural effusion
* CNS metastases by head CT scan or MRI within the past 4 weeks
* Pregnant or breast-feeding
* Prior chemotherapy or monoclonal antibodies for other cancers within 5 years prior to registration
* Prior chemotherapy for lung cancer
* Prior chest radiotherapy
* Ongoing (lasting > 14 days) or active infection or ongoing (lasting > 14 days) fever within the past 6 months
* Gross hemoptysis ≥ grade 2 (defined as ≥ ½ teaspoon of bright red blood per episode) within the past 3 months
* Bleeding ≥ grade 2 or any bleeding requiring intervention
* Clinically significant cardiovascular disease
* Myocardial infarction within the past 6 months
* New York Heart Association class III-IV congestive heart failure
* Unstable angina pectoris
* Serious cardiac arrhythmia requiring medication within the past 4 weeks
* History of hypertensive crisis or hypertensive encephalopathy
* Stroke or transient ischemic attack within the past 6 months
* Peripheral vascular disease ≥ grade 2 within the past 6 months
* Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* Psychiatric illness or social situation that would limit compliance with study requirements
* History of uncontrolled hypertension (i.e., blood pressure ≥ 150/100 mm Hg) while on stable regimen of antihypertensive therapy
* Significant traumatic injury or serious non-healing wound, ulcer, or bone fracture within the past 4 weeks
* Concurrent major surgical procedure
* Having anticipated major surgical procedure(s) during the course of the study
* Concurrent daily aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory agents (NSAIDs) known to inhibit platelet function
* Recognized immunodeficiency disease, including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia, or hereditary or congenital immunodeficiencies
* Pre-existing medical condition requiring chronic steroids or immunosuppressive therapy
* Autoimmune disease
* Known hepatitis B or C
* Immunotherapy (e.g., interferon, interleukin, sargramostim [GM-CSF], or filgrastim [G-CSF]) within 28 days prior to registration
* Prior splenectomy
* Hypersensitivity to any component of bevacizumab
* Prior core biopsy or any other minor surgical procedure, excluding the placement of a vascular access device, within 7 days prior to registration

Step 2 Inclusion Criteria:

* Serum creatinine ≤ 1.5 mg/ml or calculated creatinine clearance ≥ 45 ml/min
* Urine dipstick must be ≤ 0-1+. If urine dipstick results > 1+, 24 hour urine for protein must be obtained. Patients must have < 1g protein/24 hours to participate in the study
* Patient must be registered to step 2 within 28 days of completion of consolidation chemotherapy
* Patient must have met all eligibility requirements for Step 1
* Platelets ≥ 100,000/mm3

Step 2 Exclusion Criteria:

* Progressive disease or unevaluable disease per RECIST criteria upon post- consolidation chemotherapy evaluation
* Autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti D. Patel, Study Chair — Robert H. Lurie Cancer Center
Locations (88):
- United States (88):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford Cancer Center, Stanford, California
  - Medical Center of Central Georgia, Macon, Georgia
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Tufts Medical Center Cancer Center, Boston, Massachusetts
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: E6508 was activated on December 22, 2010, accrued its first patient on January 17, 2011, suspended per protocol on January 12, 2012 for interim toxicity analysis. The study was then reactivated on October 9, 2012 to stage 2 accrual and closed to accrual on October 13, 2014.
Period: Step 1 - Chemo RT/Consolidation Chemo
Arm/Group | Tecemotide/Bevacizumab After Chemoradiation
Started | 70
Started Treatment | 68
Completed | 39
Not Completed | 31
Not completed — Adverse Event | 10
Not completed — Death | 2
Not completed — Withdrawal by Subject | 3
Not completed — Progressive disease | 11
Not completed — Complicating disease | 1
Not completed — No show/Patient moved | 2
Not completed — Never started therapy | 2
Period: Step 2 - Maintenance Therapy
Arm/Group | Tecemotide/Bevacizumab After Chemoradiation
Started | 33 (Among 39 pts with tx completion, 4 did not register to step 2 and 2 had PD at the end of step 1.)
Completed | 0 (Max maintenance therapy was 34 cycles. No patients were off treatment due to completion of 34 cycles)
Not Completed | 33
Not completed — Progressive disease | 12
Not completed — Adverse Event | 13
Not completed — Death | 1
Not completed — Withdrawal by Subject | 4
Not completed — Complicating disease | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The primary objective was to determine the safety of combination therapy with chemoradiation, followed by consolidation, finally followed by tecemotide and bevacizumab for this patient population. Only patients who started step 2 protocol therapy were included in this analysis.
Groups:
- Step 2 - Maintenance Therapy: Maintenance therapy: Patients receive a single dose of cyclophosphamide IV over 15-30 minutes 3 days before the first dose of bevacizumab and BLP25 liposome vaccine. Patients then receive bevacizumab IV over 30-90 minutes on day 1 and BLP25 liposome vaccine subcutaneously on days 1, 8, and 15 of courses 1 and 2 and on day 1 of every other course beginning in course 4. Treatment repeats every 21 days for up to 34 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Step 2 - Maintenance Therapy
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 61 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Target Adverse Events for the Step 2 Treatment
Description: The study is to evaluate the safety of the combination of tecemotide immunotherapy with bevacizumab. The target adverse events for the combined treatment are as follows: grade 4-5 hemorrhage, esophagitis, fistula, platelet count decrease (thrombocytopenia), encephalitis infection, or hepatic failure episodes.
Time Frame: Assessed every 3 weeks while on treatment and up to 5 years
Population: All patients who received step 2 treatment
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Step 2 - Maintenance Therapy
Number analyzed (Participants) | 33
proportion of participants | 0.03 [0.003 to 0.113]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the study registration until death from any cause. Patients who were alive or lost to follow-up at the time of analysis were censored at date last known alive.
Time Frame: Every 3 months for patients < 2 years from study entry, and every 6 months if patient is 2-5 years from study entry; up to 5 years
Population: Only eligible and treated patients are included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Step 2 - Maintenance Therapy
Number analyzed (Participants) | 32
months | 42.7 [21.7 to 63.3]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from study registration to disease progression or death from any cause, whichever came first. If date of death was greater than 3 months after date of last disease assessment that showed progression-free, the patient was censored at the time of last disease assessment. Patients alive and without documented progression were censored at the date last known progression-free.
  Progression is defined using Response Evaluation Criteria In Solid Tumors (RECIST) Criteria (version 1.1), as at least 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, the appearance of new lesions, or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: Only eligible and treated patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Step 2 - Maintenance Therapy
Number analyzed (Participants) | 32
months | 14.9 [11.0 to 20.9]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment, up to 5 years
Groups:
- Step 1 - Chemoradiation and Consolidation Chemotherapy: Chemoradiotherapy: Patients receive paclitaxel intravenously (IV) over 1 hour and carboplatin IV over 15-30 minutes once a week for 6 weeks. Patients also undergo concurrent definitive radiotherapy 5 days a week for 6½ weeks. Patients with complete response (CR), partial response (PR), or stable disease (SD) proceed to consolidation chemotherapy.
  Consolidation chemotherapy: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 15-30 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with CR, PR, or SD proceed to maintenance therapy.
Arm/Group | Step 1 - Chemoradiation and Consolidation Chemotherapy | Step 2 - Maintenance Therapy
All-Cause Mortality (participants affected / at risk) | 48/68 | 21/33
Serious Adverse Events (participants affected / at risk) | 39/68 | 11/33
Other Adverse Events (participants affected / at risk) | 65/68 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 - Chemoradiation and Consolidation Chemotherapy (N=68) | Step 2 - Maintenance Therapy (N=33)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Esophageal ulcer (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 3 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 7 | 1
Neutrophil count decreased (Investigations) | 11 | 0
Platelet count decreased (Investigations) | 3 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 14 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 6
Hypotension (Vascular disorders) | 2 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 - Chemoradiation and Consolidation Chemotherapy (N=68) | Step 2 - Maintenance Therapy (N=33)
Anemia (Blood and lymphatic system disorders) | 39 | 18
Chills (General disorders) | 5 | 4
Fatigue (General disorders) | 50 | 26
Fever (General disorders) | 4 | 0
Flu like symptoms (General disorders) | 0 | 4
Injection site reaction (General disorders) | 0 | 2
Pain (General disorders) | 6 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 2
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 14 | 2
Diarrhea (Gastrointestinal disorders) | 15 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 9 | 2
Dysphagia (Gastrointestinal disorders) | 15 | 3
Esophagitis (Gastrointestinal disorders) | 32 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Mucositis oral (Gastrointestinal disorders) | 12 | 2
Nausea (Gastrointestinal disorders) | 40 | 10
Vomiting (Gastrointestinal disorders) | 13 | 3
Allergic reaction (Immune system disorders) | 4 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 13 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 3
Lymphocyte count decreased (Investigations) | 8 | 9
Neutrophil count decreased (Investigations) | 21 | 0
Platelet count decreased (Investigations) | 26 | 6
Weight loss (Investigations) | 16 | 4
White blood cell decreased (Investigations) | 40 | 10
Anorexia (Metabolism and nutrition disorders) | 14 | 9
Dehydration (Metabolism and nutrition disorders) | 6 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 3
Hypokalemia (Metabolism and nutrition disorders) | 7 | 3
Hyponatremia (Metabolism and nutrition disorders) | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 2
Dizziness (Nervous system disorders) | 4 | 3
Dysgeusia (Nervous system disorders) | 20 | 8
Headache (Nervous system disorders) | 7 | 2
Peripheral motor neuropathy (Nervous system disorders) | 12 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 22 | 17
Insomnia (Psychiatric disorders) | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory thoracic mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 6
Flushing (Vascular disorders) | 4 | 3
Hypertension (Vascular disorders) | 6 | 12
Hypotension (Vascular disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT00828009/Prot_SAP_000.pdf